CLINICAL TRIAL: NCT07220460
Title: Multicenter, Open-label Study to Evaluate the Long-term Safety and Tolerability of ABBV-932 in Subjects With Depressive Episodes Associated With Bipolar I or II Disorder
Brief Title: Study to Assess the Adverse Events of Oral ABBV-932 in Adult Participants With Depressive Episodes Associated With Bipolar I or II Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M25-456
Record Dates: First submitted 2025-09-26; First posted 2025-10-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Bipolar I or II Disorder
Keywords: Bipolar I or II Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ABBV-932 (Experimental): Participants will receive oral ABBV-932 for a 26-week treatment period followed by a 30-day follow-up
  Interventions: Drug: ABBV-932

INTERVENTIONS:
Drug: ABBV-932 — Oral Capsule

SUMMARY:
Bipolar disorder is a severe chronic mood disorder that affects up to 4% of the adult population in the United States. The purpose of this study is to assess how safe and effective ABBV-932 is in treating participants with depressive episodes associated with bipolar I or II disorder.

ABBV-932 is an investigational drug being developed for the treatment of depressive episodes in adult participants with bipolar I or II disorder. Participants with bipolar I or II disorder who are currently experiencing a depressive episode will enter the study and be treated with open-label ABBV-932. Approximately 200 adult participants with bipolar I or II disorder will be enrolled in approximately 50 sites in the United States and Puerto Rico.

Participants will receive oral capsules of ABBV-932 for a 26-week treatment period. The treatment period will be followed by a safety follow-up (SFU) period of 30 days.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regularly scheduled visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) ≥ 18.0 to ≤ 40.0 kg/m^2, inclusive.
* Participants who currently meet the Diagnostic and Statistical Manual of Mental Disorders treatment (DSM-5-TR) criteria for bipolar I or II disorder without psychotic features based on the Mini International Neuropsychiatric Interview (MINI 7.0.2), currently experiencing a depressive episode of at least 4 weeks and not exceeding 12 months.
* Normal physical examination findings, clinical laboratory test results, vital signs, and 12-lead ECG results at screening or abnormal results that are judged not clinically significant by the investigator and documented as such in the eCRF
* Participant with the following psychiatric history:

  * No history of psychiatric hospitalization (inpatient or intensive outpatient) in the past 3 months prior to screening.
  * No lifetime history of schizophrenia, other psychotic disorders, dissociative disorders, or neurocognitive disorders.
  * No history of moderate or severe substance use disorder (except nicotine) in the past 6 months prior to screening.

Exclusion Criteria:

* A total score greater than 12 on the Young Mania Rating Scale (YMRS) at baseline.
* History of an allergic reaction or significant sensitivity to constituents of the study drug (and its excipients) and/or other products in the same class.
* A concurrent medical condition that might interfere with the conduct of the study, confound the interpretation of the study results, or endanger the subject's well-being. This includes any unstable condition, history or evidence of malignancy (other than treated basal or squamous cell carcinoma), or any significant hematologic, endocrine, cardiovascular, respiratory, renal impairment or disease (subjects with eGFR < 30 mL/min), hepatic (including history of severe hepatic impairment), gastrointestinal, or neurological disorder (if there is a history of such disease but the condition has been stable for more than 1 year, does not require treatment with prohibited medications, and is judged by the investigator not to interfere with participation in the study, the subject may be included in the study).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events | Up to approximately 29 weeks
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.
Number of Participants with Abnormal Change From Baseline in Vital Sign Measurements | Up to week 26
  Number of participants with abnormal change from baseline in vital sign measurements like systolic and diastolic blood pressure will be assessed.
Number of Participants with Change from Baseline in Electrocardiogram (ECG) | Up to week 26
  12-lead resting ECG will be recorded.
Number of Participants with Abnormal Change in Clinical Laboratory Test Results Like Hematology will be Assessed | Up to week 26
  Number of participants with abnormal change in clinical laboratory test results like hematology will be assessed.
Change From Baseline in Simpson-Angus Scale (SAS) | Up to week 26
  SAS (Simpson-Angus Scale): is a 10-item rating scale for assessment of antipsychotic-induced parkinsonism in both clinical practice and research settings. Minimum: 0 (no symptoms) Maximum: 40 (very severe symptoms; 10 items scored 0-4 each).
Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) | Up to week 26
  AIMS (Abnormal Involuntary Movement Scale): assesses abnormal involuntary movements, such as tardive dyskinesia, associated with antipsychotic drugs; it measures facial, oral, extremities, and trunk movements, as well as the participant's awareness of abnormal movements. Minimum: 0 (no abnormal movements) Maximum: 42 (most severe; 7 items scored 0-4 each), some versions use 0-4 on 10 items for a max of 40/40.
Change From Baseline in Barnes Akathisia Rating Scale (BARS) | Up to week 26
  BARS (Barnes Akathisia Rating Scale): is a 4-item rating scale used to assess drug-induced akathisia. The scale comprises items for rating the observable restless movements that characterize the condition, the subjective awareness of restlessness, and any distress associated with the akathisia. Minimum: 0 (no akathisia) Maximum: 14 (severe akathisia; 4 items scored, most items 0-3 or 0-5)
Change from Baseline in Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to week 26
  C-SSRS rates an individual's degree of suicidal ideation (SI) and behaviors on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent."
Change From Baseline in the Epworth Sleepiness Scale (ESS) | Up to week 26
  ESS (Epworth Sleepiness Scale): is a scale that is intended to measure daytime sleepiness. Minimum: 0 (no sleepiness) Maximum: 24 (severe sleepiness; 8 items scored 0-3 each)
Change From Baseline in the Young Mania Rating Scale (YMRS) | Up to week 26
  The YMRS (Young Mania Rating Scale): is an 11-item, clinician-rated scale that assesses manic symptoms based on the participant's perception of their condition over the previous 48 hours, as well as the physician's clinical observations during the interview. Minimum: 0 (no mania) Maximum: 60 (severe mania; 11 items, some scored 0-4, others 0-8)
Number of Participants with Abnormal Change in Ocular Examination | Up to week 26
  Number of participants with abnormal change in ocular examinations in areas like best corrected visual acuity (BCVA), and refraction.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (41):
- United States (39):
  - Ima Clinical Research Phoenix (Alea) /ID# 278047, Phoenix, Arizona
  - Advanced Research Center /ID# 273474, Anaheim, California
  - Axiom Research /ID# 273482, Colton, California
  - Collaborative Neuroscience Research - Garden Grove /ID# 273492, Garden Grove, California
  - Sun Valley Research Center /ID# 273472, Imperial, California
  - Synergy San Diego /ID# 278340, Lemon Grove, California
  - Alliance for Research Alliance for Wellness /ID# 273477, Long Beach, California
  - Nrc Research Institute - Los Angeles /ID# 278450, Los Angeles, California
  - Excell Research /ID# 273483, Oceanside, California
  - Inland Psychiatric Medical Group Inc. /ID# 273471, Temecula, California
  - Sunwise Clinical Research /ID# 278165, Walnut Creek, California
  - Connecticut Clinical Research - Cromwell /ID# 278116, Cromwell, Connecticut
  - Cns Healthcare - Jacksonville /ID# 278332, Jacksonville, Florida
  - GMI Florida - Central Miami Medical Institute /ID# 273486, Miami, Florida
  - Allied Biomedical Res Inst Inc /ID# 273476, Miami, Florida
  - Floridian Clinical Research - Miami Lakes /ID# 279379, Miami Lakes, Florida
  - K2 Medical Research - Orlando - South Orlando Avenue /ID# 273487, Orlando, Florida
  - Apg Research /ID# 278439, Orlando, Florida
  - Segal Trials - West Broward Outpatient Research Site /ID# 273496, Tamarac, Florida
  - Atlanta Center for Medical Research /ID# 278827, Atlanta, Georgia
  - Benchmark Research /ID# 273490, Shreveport, Louisiana
  - Elixia, LLC /ID# 278446, Springfield, Massachusetts
  - Arch Clinical Trials /ID# 273481, St Louis, Missouri
  - Ima Clinical Research Las Vegas (Altea) /ID# 278054, Las Vegas, Nevada
  - Bio Behavioral Health /ID# 273478, Toms River, New Jersey
  - Integrative Clinical Trials /ID# 278040, Brooklyn, New York
  - Neurobehavioral Research /ID# 273470, Cedarhurst, New York
  - New Hope Clinical Research - Inpatient unit /ID# 273468, Charlotte, North Carolina
  - Quest Therapeutics of Avon Lake /ID# 273484, Avon Lake, Ohio
  - OSU Psychiatry Department /ID# 273495, Columbus, Ohio
  - Sooner Clinical Research /ID# 273491, Oklahoma City, Oklahoma
  - Summit Research Network - Portland - Northwest Vaughn Street /ID# 278084, Portland, Oregon
  - Lehigh Center for Clinical Research /ID# 273466, Allentown, Pennsylvania
  - FutureSearch Trials of Dallas /ID# 273473, Dallas, Texas
  - Epic Medical Research - DeSoto /ID# 278045, DeSoto, Texas
  - Perceptive Pharma Research /ID# 273485, Richmond, Texas
  - Family Psychiatry Of The Woodlands /ID# 278050, The Woodlands, Texas
  - Northwest Clinical Research Center /ID# 273480, Bellevue, Washington
  - Core Clinical Research /ID# 273498, Everett, Washington
- Puerto Rico (2):
  - INSPIRA Clinical Research /ID# 274670, San Juan
  - BDH Research /ID# 274677, San Juan

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-456